CLINICAL TRIAL: NCT04348981
Title: Preventing Cardiac Surgery Readmission With Patient Activity Tracking Technology
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding, lack of support (time)
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Dirk Varelmann, MD, Staff Anesthesiologist, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2020P000327
Record Dates: First submitted 2020-04-13; First posted 2020-04-16 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Surgery; Enhanced Recovery
Keywords: Enhanced Recovery; Cardiac Surgery; Elective; wearable; activity; readmission
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Wearable (Experimental): All patients eligible to enroll in the Enhanced Recovery after Cardiac Surgery pathway will be offered a wearable fitness tracking device.
  Interventions: Device: Wearable fitness tracking device

INTERVENTIONS:
Device: Wearable fitness tracking device — Patients having a wearable fitness tracking device will be monitored for their level of activity after surgery. Declines in activity level will prompt a phone call from the surgical provider.

SUMMARY:
The aim of this study is to detect decreased patient activity level after discharge after cardiac surgery to prevent readmissions.

Cardiac surgery is associated with a high chance of readmission within 30 days, common reasons being volume overload, arrhythmia, pulmonary complications, and infections. A decreased activity level often precedes those complications. Measuring patient activity levels using wearable activity trackers (Fitbit) may detect complications early and prompts the surgical team to contact the patient before a visit to the Emergency Room is warranted.

DETAILED DESCRIPTION:
Patients undergoing cardiac surgery are either discharged home (+/- visiting nurse), to a skilled nursing facility, or to a rehabilitation center.

Readmission rates within 30 days of cardiac surgery are ranging between 8 and 21% in the adult population (1, 2); the largest 10-center study including 5,059 patients reported a readmission rate of 19%, which is in line with the readmission rate for the Department of Cardiac Surgery at the Brigham and Women's Hospital (3). The most common causes for readmissions are volume overload/heart failure, arrhythmia, and infection (3, 4). The Centers of Medicare and Medicaid Services Readmissions Reduction Program initiated revenue penalties for an excess 30-day readmission rate [https://www.cms.gov/medicare/medicare-fee-for-service-payment/acuteinpatientpps/readmissions-reduction-program.html]. Home visits of cardiac patients after surgery on postdischarge days 2 and 5 by physician assistants had been shown to decrease readmission rate by 41%, resulting in significant cost savings ($39 saved for every $1 spent) with a readmission cost between $39,100 and $56,600 (5).

Volume overload, congestive heart failure, and infections lead to a decline in activity status. However, when assessing activity levels, self-reported data is often inaccurate and wearable devices greatly improve distinction between physical activity and sedentary time (6, 7). We therefore seek to implement data from wearable devices from patients discharge home after cardiac surgery into the software (recoupERAS) used for our Enhanced Recovery after Cardiac Surgery (ERAS cardiac surgery) program. This would allow us to non-invasively follow the patient's activity level without relying on self-reported data. We would follow the data from the hospital supplied wearable device for 30 days after cardiac surgery. In case of a decline of physical activity which would be seen in recoupERAS, we would proactively contact the patient. This would allow us to make either recommendations over the phone or invite the patient back to the cardiac surgery offices for further assessment before the patient's health status deteriorates to a point where an Emergency Department visit is necessary.

SUBJECT SELECTION All patients undergoing cardiac surgery at the Brigham and Women's Hospital (BWH) who agree to use the RecoupERAS software on their mobile device will be offered a wearable device at no cost to the patient.

a) Inclusion/Exclusion criteria:

Inclusion:

1. Patients undergoing cardiac surgery participating under the ERAS cardiac surgery protocol using the RecoupERAS software.

Exclusion:

1. Patient refusal of device
2. Patients with skin reactions to wearable devices (contact dermatitis)

IV. Subject Enrollment

1. Methods of Enrollment Patients who are undergoing cardiac surgery will be identified by the cardiac surgeon for eligibility to be enrolled in the ERAS cardiac surgery pathway. All cardiac surgery patients are seen in the BWH Weiner Center for Preoperative Evaluation. Patient enrolled into the ERAS pathway receive additional teaching, which includes the use of the RecoupERAS software, which is accessible through the patients' mobile devices. Patients will be offered a wearable device (Fitbit Charge 3), that transmits activity data to the RecoupERAS software. The patient will receive a recruitment letter and a consent form in advance of their hospital admission. The study staff will introduce the study to ensure that the patient arriving on the day of surgery has had >24hrs for consideration to participate.

   Consent will be obtained by one of the licensed physician co-investigators at the earliest opportunity after arrival in the pre-operative area. No passive recruitment methods (newspapers, advertisement, or flyers) will be used. Subjects unable to give consent themselves will not be approached for participation.
2. Procedures for obtaining informed consent (including timing of consent process) If the patient agrees to participate, a written informed consent will be obtained and a standard consent form for research approved by the IRB will be used. Any patient can withdraw from the study at any time. If the patient withdraws after receiving the wearable device, the device remains with the patient or can be send back to the study investigator for disposal.
3. Treatment assignments and randomization (if applicable) Patients who agree to participate in the study, will be equipped with a wearable fitness tracking device (Fitbit Charge 3) after surgery, either immediately before or after discharge from the ICU. The randomization is planned, the primary and secondary outcomes will be compared to a historical control group of ERAS patients.

STUDY PROCEDURES

a. Data to be collected and when the data is to be collected Basic demographic data (age, height, weight), medical condition, procedure, ICU data (intubation time, length of ICU stay), general ward data (length of hospital stay, activity data, medication) will be collected during the patients' stay as part of clinical routine and can be extracted from the electronic medical record (EMR).

Predicted morbidity, mortality, morbidity&mortality, risk of development of renal failure, predicted readmission rate, predicted risk of atrial fibrillation are collected routine as mandated by the Society of Thoracic Surgery and will be used for compare the actual complication rate to the predicted complication rate.

The wearable device will be given to the patient when he/she is being actively mobilized, either in the ICU or the general hospital ward. Data recorded by the wearable device are: steps, heart rate, sleep, estimation of calories burned, stairs, active minutes. This data is collected continuously, The RecoupERAS software will compare the data from each day to the previous one. If RecoupERAS detects a drop in active minutes, steps, or calories burned of >20%, it will prompt the provider (PA, cardiac surgery fellow, attending surgeon) to contact the patient.

1. Nabagiez JP, Shariff MA, Khan MA, et al.: Physician assistant home visit program to reduce hospital readmissions. J Thorac Cardiovasc Surg 2013; 145:225-31- 233- discussion 232-3
2. Hannan EL, Zhong Y, Lahey SJ, et al.: 30-day readmissions after coronary artery bypass graft surgery in New York State. JACC Cardiovasc Interv 2011; 4:569-576
3. Iribarne A, Chang H, Alexander JH, et al.: Readmissions after cardiac surgery: experience of the National Institutes of Health/Canadian Institutes of Health research cardiothoracic surgical trials network. Ann Thorac Surg 2014; 98:1274-1280
4. Redžek A, Mironicki M, Gvozdenović A, et al.: Predictors for hospital readmission after cardiac surgery. J Card Surg 2015; 30:1-6
5. Nabagiez JP, Shariff MA, Molloy WJ, et al.: Cost Analysis of Physician Assistant Home Visit Program to Reduce Readmissions After Cardiac Surgery. Ann Thorac Surg 2016; 102:696-702
6. Dohrn I-M, Sjöström M, Kwak L, et al.: Accelerometer-measured sedentary time and physical activity-A 15 year follow-up of mortality in a Swedish population-based cohort. Journal of Science and Medicine in Sport 2017; 1-6
7. Lee I-M, Shiroma EJ, Evenson KR, et al.: Accelerometer-Measured Physical Activity and Sedentary Behavior in Relation to All-Cause Mortality: The Women's Health Study. Circulation 2017;

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing cardiac surgery participating under the ERAS cardiac surgery protocol

Exclusion Criteria:

* Patient refusal of device
* Patients with skin reactions to wearable devices (contact dermatitis)
* upper extremity swelling
* upper extremity deep vein thrombosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Readmission | 30 days after surgery
  decreased level of activity may precede readmission

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Varelmann, MD, Principal Investigator — Brigham and Women's Hospital